CLINICAL TRIAL: NCT00328341
Title: The Use of Tissue Oxygen Monitoring in Critically Injured Patients
Status: Terminated | Type: Observational
Why Stopped: Slow to enroll.
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H6693-19472-05
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Traumatic Brain Injury; Hemorrhagic Shock; Trauma
Keywords: traumatic brain injury; hemorrhagic shock; multisystem trauma; under resuscitation; tissue oxygen monitoring
MeSH Terms: conditions — Brain Injuries, Traumatic; Shock, Hemorrhagic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is anticipated that the use of tissue oxygen monitoring to measure brain tissue oxygen and deltoid muscle oxygen will provide more precise information about focal brain ischemia and systemic hypoperfusion than current techniques and measures such as blood pressure, heart rate and intracranial pressure. Understanding the relationship between tissue oxygen tension collected from the brain and deltoid muscle in critically injured patients could lead to a broader understanding of the important metabolic and cellular events that occur following severe injury and the changes induced by therapeutic interventions. Furthermore, the use of interventions designed to improve tissue hypoxia, as measured by low brain or muscle tissue oxygen, may improve mortality or neurological recovery after systemic trauma or head trauma compared to current approaches that do not involve tissue metabolic monitoring.

DETAILED DESCRIPTION:
This is a prospective, observational, cohort study designed to investigate metabolic changes in the brain and deltoid muscle of injured patients. Study objectives are as follows:

* To establish critical, abnormal levels of tissue oxygen in the brain (PbrO2) and muscle (PmO2) of injured patients.
* To correlate PbrO2 with other currently available diagnostic measures used in head-injured patients, including ICP, mean arterial blood pressure (MAP), CPP, SjO2, CT findings, neurological examinations, and clinical outcomes from traumatic brain injury.
* To correlate PmO2 with base deficit measurements, standard physiologic variables, near infra-red oxygen levels, infectious complications, and outcomes in critically injured patients.

Investigators will enroll patients with multisystem trauma including brain injury. In addition to the results obtained from oxygen monitoring, other data collected prospectively will include:

1. Baseline Characteristics- mechanism of injury, arrival blood pressure and GCS, results of imaging procedures, age, gender, blood gas analysis, injuries and injury severity, and all operative procedures,
2. ICU Care - MAP, ICP, CPP, base deficit, oxygen saturation, CVP, cardiac output, GCS scores, short-term outcome data, infectious complications and organ dysfunction.

All physiological data will be downloaded automatically and continuously from the bedside monitor, ventilator, and oxygen monitors via a study-dedicated computer and customized software (Aristein Bioinformatics, Palo Alto, CA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Intubated and assisted mechanical ventilation
* Traumatic brain injury requiring advanced neuromonitoring
* Abbreviated injury scale 3 or more in torso. abdomen, or extremities

Exclusion Criteria:

* Age less than 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Age 18 years and older
  * Intubated and assisted mechanical ventilation
  * Traumatic brain injury requiring advanced neuromonitoring
  * Abbreviated injury scale 3 or more in torso. abdomen, or extremities
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey T Manley, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco General Hospital, San Francisco, California, United States